CLINICAL TRIAL: NCT01906463
Title: Social and Prognostic Inequalities in Patients Hospitalised for Cerebrovascular Accident (CVA) in Four Contrasting French Departments: Côte d'Or, Martinique, Guadeloupe and French Guyana Analysis of Their Impact on Vascular Risk Factors and the Management of CVA
Brief Title: Social and Prognostic Inequalities in Patients Hospitalised for Cerebrovascular Accident (CVA) in Four Contrasting French Departments
Acronym: INDIA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: bonithon PHRC N 2010
Record Dates: First submitted 2013-07-12; First posted 2013-07-24 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Symptomatic CVA (de Novo CVA)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study should also raise questions about the interest and feasibility of establishing a permanent registry of CVA in the Antilles and Guyana. Indeed in coming decades, the expected doubling of the population of persons aged over 60 years and the foreseeable changes in lifestyle will increase the burden of this disease, in particular since the region is marked by a high prevalence of arterial hypertension and diabetes and a high level of precarity. In addition, this study will provide epidemiological information on CVA, its risk factors and management, which are non-existent for the department of French Guyana where the health environment is manifestly insufficient. These data should make it possible to better evaluate the resources available and the healthcare needs in Guyana.

ELIGIBILITY:
Inclusion Criteria:

* Pre- inclusion
* Patients who have received information about the study (directly or via a person of trust),
* Patients aged more than 18 years,
* Patient hospitalised for a suspected first symptomatic CVA (whatever the mechanism), preceded or not by a transient ischemic attack (TIA),
* Patients with a cerebral imaging examination (CT-scan and/or MRI),
* in Guyana, suspicion of a first CVA according to WHO clinical criteria and who died before the authorised images for descriptive purposes,
* Patients able to answer questions personally or through a parent or a person of trust.

Definitive inclusion

- Patients with confirmed CVA diagnosed according to clinical criteria (WHO criteria) and imaging criteria.

Exclusion Criteria:

* - Patients who refuse to take part in the study,
* Patients with prior symptomatic CVA,
* Patients without cerebral imaging (except in Guyana, for patients with suspected CVA who died before imaging),
* Patients with another severe evolutive disease that could cause death in the weeks following the CVA,
* Patients who cannot be contacted by telephone at 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient from CHU Dijon , CHU Point-à-Pitre and CHU Fort-de-France,CHU Guyane
Sampling Method: Non-Probability Sample
Enrollment: 1612 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Medical history | Baseline

SECONDARY OUTCOMES:
Follow-up questionnaire: functional handicap, intercurrent hospitalisation, vital status | Month 6
Follow-up questionnaire: functional handicap, intercurrent hospitalisation, vital status | Month 1
Follow-up questionnaire: functional handicap, intercurrent hospitalisation, vital status | Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France